CLINICAL TRIAL: NCT00833040
Title: A Multicenter, Randomized, Placebo-Controlled, Crossover Study for the Evaluation of the Safety, Tolerability, and Efficacy of ARX-F02 Compared to Placebo in the Treatment of Cancer Breakthrough Pain
Brief Title: A Study for the Evaluation of the Safety, Tolerability, and Efficacy of ARX-F02 (Sufentanil NanoTab) Compared to Placebo in the Treatment of Cancer Breakthrough Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Talphera, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARX-C-003
Record Dates: First submitted 2009-01-28; First posted 2009-01-30 (Estimated); Results first posted 2015-01-01 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Cancer; Pain
Keywords: Cancer breakthrough pain
MeSH Terms: conditions — Neoplasms; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Titration of sufentanil, the DBL sufentanil & PBO (Experimental): During the Titration Phase, patients titrated to the effective dosage of sublingual sufentanil NanoTab™(20, 30, 40, 60 or 80 mcg). One sublingual sufentanil NanoTab™ was taken as needed for breakthrough pain.
  During the Double-Blind Phase, patients were then randomized to one of six treatment sequences, each of which included seven active doses of sublingual sufentanil (dosage determined in Titration Phase) and three placebo doses taken in random order. One NanoTab™ was taken as needed for breakthrough pain.
  Interventions: Drug: Sublingual sufentanil NanoTabs™ and placebo NanoTabs™

INTERVENTIONS:
Drug: Sublingual sufentanil NanoTabs™ and placebo NanoTabs™ — During the Titration Phase, patients titrated to the dose of sufentanil that provided adequate pain relief without intolerable side effects. Dosages were 20, 30, 40, 60 and 80 mcg. During the Double Blind Phase, patients were randomized to one of six sequences and took 7 doses of sufentanil (dosage determined in the titration phase, and 3 doses of placebo.
  Other Names: (ARX-F02)

SUMMARY:
The purpose of this research study was to evaluate ARX-F02 (Sufentanil NanoTab) versus placebo ("sugar" pill or inactive substance) in the management of breakthrough pain in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older with documented clinical history or evidence of a malignancy.
2. Patients must have sufficient pain to require at least the equivalent of 60 mg/day oral morphine, at least 25 mcg/hr transdermal fentanyl, at least 30 mg/day oxycodone, at least 8 mg/day oral hydromorphone for a week or longer.
3. Patient is experiencing 1 - 4 episodes of cancer breakthrough pain per day, on average but not necessarily every day, requiring use of an additional opioid analgesic.
4. Patient has a life expectancy of at least 3 months.
5. Patient must have an Eastern Cooperative Oncology Group (ECOG) performance status rating < 2.
6. Patient must be able to provide reliable documentation of pain intensity, pain relief, use of rescue medication, and global evaluation of treatment personally or with the help of a caregiver.
7. Patient must be able to enter simple commands on a Palm Pilot device, personally or with the help of a caregiver.
8. If patient is female and of childbearing potential she must have a negative urine pregnancy test at screening, and must use medically acceptable methods of birth control. Acceptable methods of birth control include oral or transdermal contraceptives, condom, spermicidal foam, IUD, progestin implant or injection, abstinence, vaginal ring, or sterilization of partner. The reason for non-childbearing potential, such as bilateral tubal ligation, bilateral oophorectomy, hysterectomy, or 1 year or more postmenopausal must be specified in the patient's CRF.
9. Patient must demonstrate the dexterity to handle the single-dose applicator that will be used for placing the NanoTab™ under the tongue.
10. Patient and/or caregiver must demonstrate ability to use the NanoTab™ retrieval tool.
11. There must be a caregiver in the home (or hospice) who will be present for at least 1 hour following each dose during titration.
12. Patient must provide written informed consent.

Exclusion Criteria:

1. Patients with uncontrollable or rapidly escalating pain.
2. Patients with a history of psychiatric disease or loss of cognitive function that would prevent patient from providing reliable study documentation.
3. Patients with oral mucositis or stomatitis.
4. Patients with a history of substance abuse within the past year.
5. Patients who are using intrathecal opioids.
6. Patients with underlying pulmonary disease such as sleep apnea or chronic obstructive pulmonary disease characterized by CO2 retention that is deemed clinically significant by the investigator.
7. Patients at risk of significant bradyarrhythmia, in the opinion of the Investigator, due to underlying heart disease.
8. Patients with abnormal chemistry or hematology that are deemed by the investigator to be clinically significant. Abnormalities that are cancer related should be documented.
9. Patients with clinically significant abnormality on the Screening ECG who, in the Investigator's opinion, should not participate in the study.
10. Patients who will be receiving chemotherapy or radiation treatment during the 3-week titration phase or 3-week double-blind phase that, in the Investigator's opinion, may dramatically alter the patient's pain level or response to pain medications.
11. Patients who are taking monoamine oxidase inhibitors (MAOIs), or have taken MAOIs within 14 days prior to enrolling in the study.
12. Patients who have participated in a clinical trial of an investigational drug or device within 30 days of screening visit.
13. Patients who, in the Investigator's opinion, should not participate in the study or may not be capable of following the study schedule or procedures for any reason.
14. Patients who are employees or family members of the Investigator, study center or AcelRx.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Clinical Trials and Research Associates, Montebello, California
  - Florida Institute of Medical Research, Jacksonville, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Sarasota Pain Medicine Research, Sarasota, Florida
  - Lovelace Scientific Resources, Venice, Florida
  - Drug Studies America, Inc., Marietta, Georgia
  - Better Health Clinical Research, Inc., Newnan, Georgia
  - International Clinical Research Institute, Overland Park, Kansas
  - Willis-Knighton Pain Management Center, Shreveport, Louisiana
  - Four Seasons Hospice & Palliative Care, Flat Rock, North Carolina
  - Center for Clinical Research, Winston-Salem, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Research Concepts Ltd, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 42 patients were enrolled and entered the Titration Phase. 36 patients determined an effective dosage of sufentanil and were randomized to the Double-Blind Phase of the study. 2 patients then terminated from the study and did not take any doses after the Titration Phase. 34 patients participated in the Double-Blind Phase of the study.
Groups:
- Sequence 1: Open Label Titration Phase - Each patient determined the effective dosage of sufentanil for their pain (20, 30, 40, 60 or 80 mcg). Patients were then randomized to one of six sequences in the Double Blind Phase in which they took ten doses of study drug.
  Double-Blind Phase/Sequence 1 - Patients took a dose of study drug, as needed for breakthrough pain, as follows: placebo treatments for the 2nd, 4th, and 7th episode of breakthrough pain and ARX-F02 (sufentanil) treatments for all other episodes of breakthrough pain (dosage of sufentanil determined in the Titration Phase).
- Sequence 2: Open Label Titration Phase - Each patient determined the effective dosage of sufentanil for their pain (20, 30, 40, 60 or 80 mcg). Patients were then randomized to one of six sequences in the Double Blind Phase in which they took ten doses of study drug.
  Double-Blind Phase/Sequence 2 - Patients took a dose of study drug, as needed for breakthrough pain, as follows: placebo treatments for the 2nd, 4th, and 8th episode of breakthrough pain and ARX-F02 (sufentanil) treatments for all other episodes of breakthrough pain (dosage of sufentanil determined in the Titration Phase).
- Sequence 3: Open Label Titration Phase - Each patient determined the effective dosage of sufentanil for their pain (20, 30, 40, 60 or 80 mcg). Patients were then randomized to one of six sequences in the Double Blind Phase in which they took ten doses of study drug.
  Double-Blind Phase/Sequence 3 - Patients took a dose of study drug, as needed for breakthrough pain, as follows: placebo treatments for the 2nd, 5th, and 9th episode of breakthrough pain and ARX-F02 (sufentanil) treatments for all other episodes of breakthrough pain (dosage of sufentanil determined in the Titration Phase).
- Sequence 4: Open Label Titration Phase - Each patient determined the effective dosage of sufentanil for their pain (20, 30, 40, 60 or 80 mcg). Patients were then randomized to one of six sequences in the Double Blind Phase in which they took ten doses of study drug.
  Double-Blind Phase/Sequence 4 - Patients took a dose of study drug, as needed for breakthrough pain, as follows: placebo treatments for the 3rd, 5th, and 7th episode of breakthrough pain and ARX-F02 (sufentanil) treatments for all other episodes of breakthrough pain (dosage of sufentanil determined in the Titration Phase).
- Sequence 5: Open Label Titration Phase - Each patient determined the effective dosage of sufentanil for their pain (20, 30, 40, 60 or 80 mcg). Patients were then randomized to one of six sequences in the Double Blind Phase in which they took ten doses of study drug.
  Double-Blind Phase/Sequence 5 - Patients took a dose of study drug, as needed for breakthrough pain, as follows: placebo treatments for the 3rd, 6th, and 8th episode of breakthrough pain and ARX-F02 (sufentanil) treatments for all other episodes of breakthrough pain (dosage of sufentanil determined in the Titration Phase).
- Sequence 6: Open Label Titration Phase - Each patient determined the effective dosage of sufentanil for their pain (20, 30, 40, 60 or 80 mcg). Patients were then randomized to one of six sequences in the Double Blind Phase in which they took ten doses of study drug.
  Double-Blind Phase/Sequence 6 - Patients took a dose of study drug, as needed for breakthrough pain, as follows: placebo treatments for the 3rd, 6th, and 10th episode of breakthrough pain and ARX-F02 (sufentanil) treatments for all other episodes of breakthrough pain (dosage of sufentanil determined in the Titration Phase).
Period: Overall Study
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 6 | 6 | 6 | 6 | 5 | 5
Completed | 6 | 6 | 6 | 6 | 5 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Sufentanil Followed by Sufentanil and PBO: During the Titration Phase, patients titrated to the effective dosage of sufentanil NanoTab™(20, 30, 40, 60 or 80 mcg). One sufentanil NanoTab™ was taken as needed for breakthrough pain.
  During the Double-Blind Phase, patients were then randomized to one of six treatment sequences, each of which included seven active (dosage determined in Titration Phase) and three placebo doses taken in random order per. One NanoTab™ was taken as needed for breakthrough pain.
Arm/Group | Sufentanil Followed by Sufentanil and PBO
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted SPID30
Description: time-weighted SPID30 is the sum of the pain intensity difference (PID) over the 30 minute time period. A pain intensity score of 0 (no pain) to 10 (worse possible pain) is recorded at pre-dose, 10, 15, 30, 45, and 60 minutes post-dose. The pain score at each assessment time through 30 minutes is subtracted from the baseline pain score to provide the total sum score or SPID30. A higher SPID30 is better and indicates a reduction in pain intensity compared to the baseline score.
Time Frame: 30 minutes after dosing
Population: Intent to treat population defined as all patients who took at least one dose of study drug
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Double Blind Phase of 7 Sufentanil Tablets; Double Blind Phase of 3 Pbo Tablets: Open Label Titration Phase - Each patient determined the effective dosage of sufentanil for their pain (20, 30, 40, 60 or 80 mcg). In the Double-Blind Phase, each patient was randomized to one of six treatment sequences in which the patient took seven active sufentanil doses (dosage determined in the Titration Phase) and three placebo doses as needed for breakthrough pain.
Arm/Group | Double Blind Phase of 7 Sufentanil Tablets | Double Blind Phase of 3 Pbo Tablets
Number analyzed (Participants) | 34 | 34
units on a scale | 59.9 (6.25) | 42.6 (6.86)
Statistical Analysis 1: Comparison: Double Blind Phase of 7 Sufentanil Tablets vs Double Blind Phase of 3 Pbo Tablets; difference between the active and placebo groups; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 17.3, Standard Error of Mean 4.49

ADVERSE EVENTS:
Time Frame: The length of the study varied for each patient. AEs were reported and collected during the titration period and well as the treatment period and for 12 hour after the last dose of study medication.
Groups:
- Titration of Sufentanil Followed by Sufentanil and PBO: During the Titration Phase, patients titrated to their personal effective strength of sufentanil NanoTab™(20, 30, 40, 60 or 80 mcg). One sufentanil NanoTab™ was taken for each episode of breakthrough pain.
  During the Double-Blind Phase, patients were randomized to one of six treatment sequences, each of which included seven active doses (the strength determined in Titration Phase) and three placebo doses. The ten doses were in random order. One NanoTab™ was taken for each episode of breakthrough pain.
Arm/Group | Titration of Sufentanil Followed by Sufentanil and PBO
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 1/34
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Titration of Sufentanil Followed by Sufentanil and PBO (N=34)
Aphasia (Nervous system disorders) | 1 — All adverse events related to study drug and were reported by one patient who received 40 mcg.
Decreased Cognition (Nervous system disorders) | 1
Right Hemiparesis (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Sedation (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication without prior written consent